CLINICAL TRIAL: NCT05007990
Title: Caregiving Networks Across Disease Context and the Life Course: A Comparative Longitudinal Study
Brief Title: Caregiving Networks Across Disease Context and the Life Course
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 210020; 21-HG-0020
Record Dates: First submitted 2021-08-14; First posted 2021-08-17 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09-08

CONDITIONS: Inherited Metabolic Disorders; Undiagnosed Diseases; Batten's Disease; Tay Sachs; Diabetes
Keywords: Social Support; Rare Diseases; Natural History; Genetic Conditions; Family Network
MeSH Terms: conditions — Undiagnosed Diseases; Neuronal Ceroid-Lipofuscinoses; Diabetes Mellitus; Rare Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active: Participants include individuals who are caregivers of an individual with a chronic medical condition, OR individuals who support caregivers of an individual with a chronic medical condition.
- Bereaved: Participants include individuals who were caregivers of an individual with a chronic medical condition who has died, OR individuals who support the caregiver.

SUMMARY:
Background:

In the U.S., about 53 million informal, unpaid caregivers provide care to a person who is ill, is disabled, or has age-related loss of function. These caregivers may be adult children, spouses, parents, or others. The stress of providing long-term care affects caregivers health and well-being. Researchers want to learn more about this stress and its effects.

Objective:

To learn how the caregiving process affects the health and well-being of caregivers over time.

Eligibility:

Adults aged 18 years and older who are caregivers for a person with a chronic medical condition and who have already given consent to take part in other study activities.

Design:

Participants will be put in different groups. They will complete some or all of the following tasks over 1 year. They may repeat these tasks once a year for up to 5 years.

Participants will fill out 2 online surveys. One will ask about their health and their caregiving experience. The other will ask them to list people in their social network and their care recipient s social network who give them support.

Participants will have a 2-part phone interview. It will be audio recorded. In part 1, they will be asked about the people they listed in the survey. In part 2, they will be asked about their caregiving experience and events in the care recipient s life.

Participants may fill out a weeklong diary every 3 months. It will ask about their daily social activities, well-being, and stress levels. It will also ask about their thoughts and feelings about caregiving.

Participants may give a blood sample each year they are in the study.

...

DETAILED DESCRIPTION:
Study Description: Caregivers will be invited to participate in surveys and interviews to assess their cognitions and emotions about caregiving, caregiving burden, and caregiving or support network systems during the life of the Care Recipient. The study will also include a bereavement component, in which families who have experienced the death of a Care Recipient may choose to participate. In addition, biomarkers may be evaluated in consenting individuals to assess genetic susceptibility to stress and stress-related dysregulations in the endocrine and immune systems.

Objectives: The primary objective of this study is to investigate the natural history of family caregiver stress over time, providing opportunity to understand the social, psychological, behavioral, and biological factors that characterize caregivers response to long-term caregiving during the life and after death of a Care Recipient with a chronic medical condition.

Endpoints: To assess the change over time in terms of social, psychological, behavioral, and biological factors associated with caregiving.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

* Adults aged 18 years and older
* If the Care Recipient is living, they must self-identify as a primary caregiver to the Care Recipient (individual with a chronic medical condition), OR if the Care Recipient is deceased, they must self-identify as having been a primary caregiver to the now-deceased Care Recipient, OR they must otherwise be identified (i.e., referred) by a participant as a part of the caregiving network
* Ability to consent to research
* Fluency in English will be needed to complete interview as well as to read, comprehend surveys and consent forms, as appropriate validated measures in other languages are not readily available.
* Physically capable of participating in applicable assessments

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from this study:

* Care Recipients (as defined in this protocol)
* Staff of NHGRI

Staff of NHGRI are unable to participate in this study as a safeguard against the risk of ethical concerns. As per OHSRP SOP 404, NIH staff may be a vulnerable class of study subjects. Excluding staff of the Institute conducting the study assures there will not be any perceived or actual conflict of interest, pressure/coercion to participate among co-workers, subordinates, work unit-members, etc. As further noted in OHSRP SOP 404, exclusion further protects this class of subjects privacy and confidentiality; and protects the study s scientific integrity.

Persons with impaired neuro-sensory or decision-making ability (adults unable to provide consent) will not be enrolled in the study. Persons with impaired neuro-sensory or decision making ability would not be able to participate with independent responses to the various social behavioral measures we use in the study interview and survey. Learning information about these individuals through other people instead of themselves would introduce bias to this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Referencing the enrollment numbers from the study of Inherited Diseases, Caregiving, and Social Networks (PI: Koehly, protocol #12HG0022), this longitudinal study will initially recruit from existing participants enrolled in #12HG0022. Family caregivers providing ongoing support for a chronically ill individual may be identified and informed about the Longitudinal Caregiving Study by an intramural NIH investigator involved in natural history protocols. Caregivers may also be recruited through other (nonNIH) clinicians, researchers, advocacy groups, online and traditional advertising, and ClinicalTrials.gov.
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Natural History | Annually / quarterly
  Investigate the natural history of family caregiving to identify the social, psychological, behavioral, and biological mechanisms that determine possible long-term changes in health during the life and after death of a Care Recipient with a chronic medical condition.

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Koehly, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-HG-0020.html